CLINICAL TRIAL: NCT01312064
Title: Clinical Outcome of de Novo Everolimus-based Immunosuppressive Therapy for Renal Transplantation Using Rituximab Induction
Brief Title: De Novo Everolimus-based Therapy for Renal Transplantation Using Rituximab Induction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty collecting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201011050MB
Record Dates: First submitted 2011-01-26; First posted 2011-03-10 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-11

CONDITIONS: Renal Insufficiency
Keywords: rituximab; everolimus
MeSH Terms: conditions — Renal Insufficiency | interventions — Rituximab; Everolimus; thymoglobulin; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rituximab and everolimus (Active Comparator): Patients of the study arm will receive rituximab (375mg/m2) induction and subsequently everolimus-based immunosuppressive therapy. Everolimus will be given with an initial dose of 1 mg bid within 24 hrs after reperfusion, adjusted to a target trough blood level of 6-10 ng/ml for the first 6 months after transplantation.
  Interventions: Drug: rituximab and everolimus
- thymoglobulin and tacrolimus (Active Comparator): The control arm will receive thymoglobulin induction and tacrolimus-based immunosuppressive therapy. The dose of thymoglobulin would be 1.0mg/kg/d for 3 days25. The first dose of thymoglobulin will be administered before graft kidney reperfusion, and so is rituximab. All patients will receive corticosteroid therapy as usual. The initial daily dose of tacrolimus will be 0.15 mg/kg/d given in two doses starting within 24 hours after transplantation. The doses of tacrolimus will be adjusted to target the whole blood trough levels between 8 to 12 ng/ml during the first 30 days after transplantation, and tapered to 6 to 10 ng/ml at 6 months.
  Interventions: Drug: thymoglobulin and tacrolimus

INTERVENTIONS:
Drug: rituximab and everolimus — rituximab (375mg/m2) induction and subsequently everolimus-based immunosuppressive therapy. Everolimus initial dose: 1 mg bid within 24 hrs after reperfusion, adjusted to a target trough blood level of 6-10 ng/ml for the first 6 months after transplantation.
  Other Names: mabthera
  Arms: rituximab and everolimus
Drug: thymoglobulin and tacrolimus — thymoglobulin induction and tacrolimus-based immunosuppressive therapy. thymoglobulin dose: 1.0mg/kg/d for 3 days daily dose of tacrolimus: 0.15 mg/kg/d given in two doses starting within 24 hours after transplantation
  Other Names: ATG
  Arms: thymoglobulin and tacrolimus

SUMMARY:
The investigators hypothesized that everolimus-based immunosuppressive therapy combined with rituximab induction could provide comparable safety profiles for renal transplant patients, as compared to standard immunosuppressive therapy using thymoglobulin induction, tacrolimus, mycophenolate mofetil and steroids, in terms of acute rejection rate and renal function.

Rituximab was reported to reverse refractory acute kidney transplant rejection. Combined with immunoadsorption with or without IVIG, rituximab could successfully prevent antibody-mediated rejection in ABO-incompatible renal transplantation. This study is to assess whether a CNI-free regimen including B-cell depleting antibody induction, everolimus and MMF results in comparable long-term function without a negative impact on safety or efficacy of immunosuppression. This study will be open-label and two-arm randomized (2:1).

DETAILED DESCRIPTION:
Patients of the study arm (2/3 of the patients) will receive rituximab (375mg/m2) induction and subsequently everolimus-based immunosuppressive therapy. The control arm (1/3 of the patients) will receive thymoglobulin induction and tacrolimus-based immunosuppressive therapy. Everolimus will be given with an initial dose of 1 mg bid within 24 hrs after reperfusion, adjusted to a target trough blood level of 6-10 ng/ml for the first 6 months after transplantation. The control arm (1/3 of the patients) will receive thymoglobulin induction and tacrolimus-based immunosuppressive therapy. The dose of thymoglobulin would be 1.0mg/kg/d for 3 days25. The first dose of thymoglobulin will be administered before graft kidney reperfusion, and so is rituximab. All patients will receive corticosteroid therapy as usual. The initial daily dose of tacrolimus will be 0.15 mg/kg/d given in two doses starting within 24 hours after transplantation. The doses of tacrolimus will be adjusted to target the whole blood trough levels between 8 to 12 ng/ml during the first 30 days after transplantation, and tapered to 6 to 10 ng/ml at 6 months. All patients will receive mycophenolate mofetil (MMF) starting at 2 g/d in divided doses, and then adjusted to maintain WBC between 4000~6000/mm3. All patients entering this study will receive co-trimoxazole as prophylactic medication for at least 12 weeks post-operatively. Valgancyclovir will be given for anti-viral prophylaxis. During the transplant operation, renal biopsy will be performed before vascular perfusion for baseline pathology, and a follow-up biopsy will be scheduled at 2 years after transplantation. The primary endpoint will be incidence of acute rejection, and the secondary endpoints include renal function, graft and patient survival.

Male and female adult patients who are to receive renal transplantation may enter the study. The intention is to enroll 90 patients who have fulfilled inclusion/exclusion criteria into the study. Sixty patients will receive rituximab and everolimus-based therapy, but the other thirty patients will receive thymoglobulin and tacrolimus-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at 15-65 years of age undergoing renal transplantation
* Patients who have been informed of the potential risks and side effects of the study
* Patients who have given written informed consent to participate in the study
* Females who are not pregnant or nursing women (pregnancy test required)

Exclusion Criteria:

* Donor age greater than 65 years
* Patients receiving a perfectly matched kidney (6 matches HLA A, B, DR)
* Patients who are recipients of multiple solid organ transplants
* Patients undergoing second or subsequent transplantation
* Patients with pre-transplant PRA > 30%
* Patients with ABO incompatibility or positive lymphocytotoxicity
* Patients with severe, active infection
* Patients who have an abnormal liver profile such as ALT, AST, alkaline phosphatase or total bilirubin >3 times the upper normal limit
* Patient who are HIV-positive or hepatitis C (PCR+ only) B surface antigen positive
* Patients who have been treated with an investigational drug or therapy within one month prior to entry or who will be so treated within 6 months of transplantation
* Patients with a history of malignancy within the last five years except excised squamous or basal cell carcinoma
* Patients with a history of alcohol or drug abuse or signs of alcohol-induced organ damage, mental dysfunction or other factors limiting their ability to comply fully with the study requirements.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
acute rejection | 6 months
  The log-rank test will be used to analyse the percentage of rejection-free survival between the two groups. Any patient with a suspicious rejection episode will reveive renal biopsy.

SECONDARY OUTCOMES:
renal function | 24 months
  Renal function will be estimated by Cockcroft-Gault formula and analysed by 2-tailed student test.
adverse event | 24 months
  All adverse events and serious adverse events, infections, and malignancies,will be regular monitored including laboratory variables and vital signs and the performance of physical examinations. Number of participants with adverse events will be compared with Chi-square tests.

CONTACTS AND LOCATIONS:
Overall Officials: MK Tsai, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan